CLINICAL TRIAL: NCT04713579
Title: Timing of Stoma Closure in Neonates (ToSCiN)
Brief Title: Timing of Stoma Closure in Neonates
Acronym: ToSCiN
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Oxford (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: B00984; G69250 (Other Grant/Funding Number: Manchester University NHS Foundation Trust)
Record Dates: First submitted 2020-11-09; First posted 2021-01-19 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Enterocolitis, Necrotizing; Atresia; Bowel; Gastroschisis; Meconium Ileus; Premature Birth; Bowel Obstruction; Perforation Bowel
Keywords: Stoma closure; Infant; Neonatal
MeSH Terms: conditions — Enterocolitis, Necrotizing; Intestinal Atresia; Gastroschisis; Meconium Ileus; Premature Birth; Intestinal Obstruction; Intestinal Perforation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premature infants: Infants born prematurely requiring a stoma for condition such as necrotizing enterocolitis (NEC) or spontaneous intestinal perforation (SIP).
  Interventions: Other: No intervention - observational study
- Term Infants: Infants born closer to term requiring a stoma e.g. for congenital causes of bowel obstruction such as intestinal atresia, gastroschisis or meconium ileus
  Interventions: Other: No intervention - observational study

INTERVENTIONS:
Other: No intervention - observational study — There is no intervention in this study as it is purely observational.

SUMMARY:
Some babies require emergency surgery on their tummy in the first few months of life. This is most commonly because they were born prematurely and developed a bowel problem (called NEC) or a blockage of the bowel. As part of this surgery, the ends of the bowel may be brought to the skin surface (called a stoma) to divert stool into a bag. The stoma allows time for the bowel to rest and recover and is intended to be temporary with reversal later on. The best time to reverse or "close" the stoma is unknown. Stomas may cause dehydration, poor growth and skin problems so earlier closure may be better; however surgery is safer when babies are older and bigger so later closure may be better.

This study aims to answer the question, 'is it feasible to conduct a clinical trial comparing 'early' vs. 'late' stoma closure in neonates?' It has a series of specific objectives which incorporate: (i) describing current UK practice; (ii) establishing whether or not a clinical trial (and exactly what form of trial) is acceptable to parents and clinicians; and (iii) establishing the design of a potential trial, including defining the intervention ('early vs. late') and the population of infants to be included, how infants should be recruited and what information should be collected (outcomes).

The investigators will ask parents and health professionals for their views and whether they would take part in a future trial and information about babies who have recently had a stoma to find out which factors influence the timing of closure. They will also analyse 6 years of data from an existing database, the National Neonatal Research Database to estimate the numbers of babies affected, understand current practice and outcomes for these babies to help decide whether a clinical trial is possible.

DETAILED DESCRIPTION:
Neonates undergoing emergency abdominal surgery frequently require stoma formation. Reversing (closing) these stomas with a second operation is an essential part of the infant's recovery. The timing of this closure is highly variable around the United Kingdom (UK) and the best time remains unclear. Current evidence is of low methodological quality and presents mixed conclusions: determining the best time has significant potential benefits for: (i) infant health outcomes (short-term e.g. avoiding complications and long-term e.g. growth and neurodevelopment); ii) families (e.g. reduced Neonatal Intensive Care Unit (NICU) stay); and iii) healthcare providers (e.g. reduced costs). Ideally, a clinical trial to compare early and late closure would be conducted but this is likely to be challenging and may not be feasible or acceptable to parents and clinicians.

Aims and objectives:

This study aims to answer the question, 'is it feasible to conduct a clinical trial comparing 'early' vs. 'late' stoma closure in neonates?' It has a series of specific objectives which incorporate: (i) describing current UK practice; (ii) establishing whether or not a clinical trial (and exactly what form of trial) is acceptable to parents and clinicians; and (iii) establishing the design of a potential trial, including defining the intervention ('early vs. late') and the population of infants to be included, how infants should be recruited and what information should be collected (outcomes).

Methods:

The study will use a mixed-methods approach comprising three parallel workstreams (WS). WS 1 will be a national survey of clinician perspectives of neonatal stoma closure. WS 2 will use an observational cohort study, interviews, questionnaires and focus groups. WS 3 will analyse three existing large databases (National Neonatal Research Database (NNRD), Health Episode Statistics (HES) and British Association of Paediatric Surgeons Congenital Anomalies Surveillance System (BAPS-CASS)).

The findings of these WS will be combined and presented at a final, trial design meeting where conclusions about trial feasibility will be reached and if appropriate, an outline of a trial protocol agreed.

Anticipated impact and dissemination:

The principal impact will be determining whether or not a definitive trial can go ahead: if the study demonstrates that a trial is feasible then the investigators will use their findings to design a trial that is acceptable to parents and clinicians; that includes the most appropriate infants; that measures outcomes important to parents and clinicians and ultimately, answers the question: when is the best time to close an infant's stoma? Findings will be disseminated at national meetings of relevant professionals, through social media (including patient groups), to funding bodies and in open access publications.

ELIGIBILITY:
Workstream 1

Inclusion criteria:

* Neonatologists in surgical NICUs, neonatal surgeons, neonatal dieticians and neonatal surgical nurses.

Workstream 2.1

Inclusion criteria:

* Infants having a stoma as part of emergency surgery before 44 weeks post-conceptual age: Group A preterm infants who have stomas formed for necrotising enterocolitis, spontaneous intestinal perforation or other intestinal pathology, and Group B infants (usually born closer to term) who have congenital anomalies that lead to bowel obstruction (e.g. intestinal atresias; meconium ileus and other conditions such as complicated gastroschisis).

Exclusion criteria:

* Cases where a stoma is part of a planned treatment pathway e.g. for an anorectal malformation or Hirschsprung's disease.
* Infants who have a stoma formed after 44 weeks post-conceptual age.

Workstream 2.2

Inclusion criteria:

* Lead surgeons and neonatologists caring for infants recruited to WS 2.1.

Workstream 2.3

Inclusion criteria:

* Parents of premature and term infants who have had an stoma in the last three years (including parents of infants recruited to WS 2.1).
* Clinicians in participating surgical units, who are involved in the treatment of infants requiring emergency stoma closure.

Exclusion criteria:

* Parents who do not speak English.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Workstream 1: clinicians involved in caring for infants with stomas in UK surgical units.
  Workstream 2.1: Infants who have had a stoma formed as part of emergency surgery before 44 weeks post-conceptual age.
  Workstream 2.2: clinicians involved in caring for infants recruited to WS 2.1.
  Workstream 2.3: Parents of premature and term infants who have had an stoma in the last three years; clinicians in participating surgical units, who are involved in the treatment of infants requiring emergency stoma closure.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of a future trial comparing early and late stoma closure | through study completion, an average of 1 year
  The key research question 'Is it feasible to conduct a clinical trial comparing 'early' vs. 'late' stoma closure in neonates?' will be answered by completing the series of secondary outcome measures using qualitative mixed research methods

SECONDARY OUTCOMES:
To establish current UK practice for stoma closure in neonates | through study completion, an average of 1 year
  Find out what is currently happening in the UK for stoma closure in babies
To determine whether there is equipoise amongst clinicians (neonatal surgeons, and neonatologists) and allied health professionals (specialist nurses and dieticians) over when it is best to close stomas in neonates | through study completion, an average of 1 year
  Find out whether surgeons, neonatal doctors and other professionals like dietitians are genuinely uncertain about when it is best for stomas to be closed
To determine the willingness of parents, neonatal surgeons and neonatologists to include neonates in a trial that would randomise to 'early' or 'late' stoma closure and identify potential barriers to recruitment. | through study completion, an average of 1 year
  Find out if parents, surgeons and neonatal doctors would be willing to include babies in a trial that would randomly allocate them (like tossing a coin) to 'early' or 'late' stoma closure
To define 'early' and 'late' stoma closure for a potential trial. | through study completion, an average of 1 year
  Decide what is meant by 'early' and 'late' stoma closure for a potential trial
Identify a group of babies for inclusion in a trial and find out how many of these babies could be included in the UK. | through study completion, an average of 1 year
  To define a population of neonates for inclusion in a trial (in whom there is significant uncertainty over timing) and determine how many babies are eligible for inclusion.
Find the most appropriate design for a potential trial | through study completion, an average of 1 year
  To establish the most appropriate design and outcome measures for a trial.
To assess the suitability of using routinely collected data for gathering clinical information for a trial. | through study completion, an average of 1 year
  Find out if current national databases could be used for gathering the required information for a potential trial

CONTACTS AND LOCATIONS:
Overall Officials: Nick Lansdale, MB FRCS PhD, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom